CLINICAL TRIAL: NCT04458311
Title: ACTION: Phase I/II Trial of Abiraterone Acetate in Combination With Tildrakizumab (Anti-IL23 Targeting Monoclonal Antibody) in Men With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: Abiraterone Acetate in Combination With Tildrakizumab
Acronym: ACTIon
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funder decided that response outcomes to date did not support continuation of the study.
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCR5163
Record Dates: First submitted 2020-06-11; First posted 2020-07-07 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
MeSH Terms: interventions — Abiraterone Acetate; tildrakizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phase I (Experimental): Increasing doses of tildrakizumab in combination with a fixed dose of abiraterone to establish the recommended phase II dose in patients with metastatic castration resistant prostate cancer..
  Interventions: Drug: Abiraterone Acetate; Drug: Tildrakizumab
- Phase II (Experimental): The Phase II part of the study will evaluate the recommended phase II dose identified in Phase I of the study in patients with metastatic castration resistant prostate cancer.
  Interventions: Drug: Abiraterone Acetate; Drug: Tildrakizumab

INTERVENTIONS:
Drug: Abiraterone Acetate — Supplied as 125 mg tablets
  Other Names: Yonsa
Drug: Tildrakizumab — Tildrakizumab will be supplied in single-use 100 mg/mL glass vials intended for IV infusion.

SUMMARY:
The purpose of this study is to find out the side effects and safety of a combination of the anti-IL23 targeting monoclonal antibody tildrakizumab in combination with abiraterone acetate in men with metastatic castration resistant prostate cancer and to determine the most appropriate dose of this combination. In the Phase I part of this study small groups of patients will be treated with increasing doses of tildrakizumab in combination with a fixed dose of abiraterone acetate (500mg once daily). Once Phase I has been completed the combination with the optimum safety and pharmacokinetic/pharmacodynamic profile will be taken forward to the Phase II part of the study. The Phase II part of the study will evaluate the optimized dose/schedule identified in Phase I of the study in patients with metastatic castration resistant prostate cancer.

DETAILED DESCRIPTION:
The trial will be divided into 2 parts: Phase I and Phase II.

The Phase I study will adopt a Bayesian Continual Reassessment Method. Patients will receive single-agent abiraterone run-in of 500 mg orally, once daily (continuous dosing) along with prednisolone at 5 mg BD until PSA progression on abiraterone monotherapy is confirmed. This run-in will not be required if patients have been treated with abiraterone in the previous 6 months. Upon confirmation of PSA progression, tildrakizumab IV will be started and given once every 4-weeks in combination with the fixed dose abiraterone (and prednisolone). The starting dose of tildrakizumab will be 100mg, with single dose escalations to 300mg and 600mg to determine the RP2D to take forward to the Phase II study. Depending on the number of responses observed, dose levels that are deemed tolerable may be expanded to up to a total of 10 patients who are evaluable for response.

The Phase II study will employ a two-stage Minimax design, recruiting up to 25 patients. During the first stage, 15 evaluable patients will be enrolled and followed for a minimum of 2 cycles each. If there are one or more responses confirmed at least 4-weeks later, an additional 10 evaluable patients will be recruited. If 4 or more responses are seen in the 25 patients evaluable for response, the combination will be deemed successful, warranting further evaluation in subsequent phases of testing. In the phase II study, patients will start taking 500mg abiraterone as an oral tablet once daily along with 5mg of prednisolone twice daily until PSA progression on abiraterone monotherapy is confirmed. This run-in will not be required if patients have been treated with abiraterone in the previous 6 months. Upon confirmation of PSA progression, the tildrakizumab will be given as an intravenous infusion at the dose established in the Phase I safety part of the study in combination with the abiraterone (and prednisolone) from combination Cycle 1 Day 1 onwards.

ELIGIBILITY:
Inclusion Criteria:

1. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up.
2. Age 18 or above.
3. Histologically or cytologically proven adenocarcinoma of the prostate.
4. Metastatic castration resistant prostate cancer
5. Documented prostate cancer progression as assessed by the investigator with RECIST (v1.1) and PCWG3 criteria with at least one of the following criteria:

   1. Progression of soft tissue/visceral disease by RECIST (v1.1) and/or,
   2. Progression of bone disease by PCWG3 bone scan criteria and/or,
   3. Progression of PSA by PCWG3 PSA criteria and/or,
   4. Clinical progression with worsening pain and need for palliative radiotherapy for bone metastases.
6. Patients that have progressed after either enzalutamide or abiraterone treatment (having received a minimum of 12-weeks of enzalutamide or abiraterone).
7. Ongoing androgen deprivation with a luteinizing hormone releasing hormone analogue (unless the patient is surgically castrated) maintaining serum testosterone of less than 50 ng/dL (less than 2.0 nM) is mandatory.
8. Life expectancy of at least 12-weeks.
9. World Health Organisation (WHO) performance status of 0-2
10. Able to swallow the study drug.
11. Archival tissue must be available for research analysis.
12. Patients must have disease that is amenable to biopsy and must be willing to undergo tumour biopsies.
13. Haematological and biochemical indices within the required ranges in protocol. These measurements must be performed within two weeks prior to the patient's first dose of any investigational medicinal products (IMP).

Exclusion Criteria:

1. Patients with predominantly small cell or neuroendocrine differentiated prostate cancer are not eligible.
2. Prior therapy, including major surgery, chemotherapy, radium-223, or other anti-cancer therapy within 4-weeks prior to IMP administration. Patients who were receiving abiraterone acetate (Zytiga® or Yonsa™) immediately prior to trial entry will not need to undergo a washout period. The use of bisphosphonates or RANK ligand inhibitors, provided the patient has been on a stable dose without any dose adjustment for at least 30 days prior to combination Cycle 1 Day 1, in patients with known osteopenia or osteoporosis or bone metastases is permitted. A single fraction of palliative radiation is permitted if at least 14-days before starting trial treatment.
3. Prior hormonal treatment exclusions as follows:

   * prior flutamide treatment during previous four-weeks N.B. Patients whose PSA did not decline in response to antiandrogens given as a second line or later intervention will only require a 14-day washout;
   * prior bicalutamide (Casodex) and nilutimide (Nilandron) treatment during previous six-weeks;
   * prior progesterone, medroxyprogesterone, progestins, cyproterone acetate, tamoxifen, and 5-alpha reductase inhibitors during previous two-weeks (14-days).
4. Live vaccine within 4 weeks of starting trial treatment and up to 17 weeks from the last dose of Tildrakizumab.
5. Prior limited field radiotherapy within the previous two weeks (14-days), or wide field radiotherapy within the previous four weeks of trial entry.
6. Participation in another interventional clinical trial and any concurrent treatment with any investigational drug within four weeks prior to IMP administration.
7. Any toxicities due to prior chemotherapy and/or radiotherapy that have not resolved to NCI-CTCAE v5.0 Grade ≤1 with the exception of chemotherapy induced alopecia and Grade 2 peripheral neuropathy.
8. Clinical evidence of hyperaldosteronism or hypopituitarism.
9. Use of drugs that are known strong CYP3A4 inducers and CYP2D6 substrates with a narrow therapeutic index (please refer to http://medicine.iupui.edu/clinpharm/ddis/table.aspx). Seville orange or grapefruit products, and any herbal medications should be avoided for four weeks prior to starting trial treatment.
10. Malabsorption syndrome or other condition that would interfere with enteral absorption of the study drugs.
11. Known intracerebral metastases
12. Any of the following cardiac criteria:

    1. QT interval > 470 msec.
    2. Clinically important abnormalities including rhythm, conduction or ECG changes (left bundle branch block, third degree heart block).
    3. Factors predisposing to QT prolongation including congenital long QT syndrome; family history of prolonged QT syndrome, unexplained sudden death (under 40); concomitant medications known to prolong QT interval.
    4. Coronary artery bypass, angioplasty, vascular stent, myocardial infarction, angina or congestive heart failure (NYHA ≥ grade 2) in the last 6 months (see the NYHA scale).
13. Uncontrolled hypotension (systolic blood pressure < 90mmHg and or diastolic blood pressure < 50 mmHg).
14. Uncontrolled hypertension on optimal medication (systolic blood pressure >180, diastolic blood pressure > 100).
15. Patients with known history of adrenal insufficiency or mineralocorticoid excess.
16. Patients with a significant history of liver disease (Child-Pugh B or C, viral or other hepatitis, current alcohol abuse or cirrhosis).
17. Known history of hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
18. At high medical risk because of non-malignant systemic disease including active infection, latent or active TB.
19. Known history of tuberculosis.
20. Poorly controlled diabetes with HbA1C > 7.5%.
21. Malignancy other than prostate cancer within three-years of trial entry with the exception of adequately treated basal cell carcinoma. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy must have no evidence of that disease for at least-three years and be deemed at negligible risk for recurrence, are deemed eligible.
22. Immunocompromised patients including patients who have previously received organ transplants or are on long-term immunosuppression (e.g. corticosteroids of > 10 mg daily equivalent of prednisolone).
23. Active or uncontrolled autoimmune disease requiring corticosteroid therapy or other forms of systemic immunosuppression.
24. Any other finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect interpretation of the results or renders the patients at high risk from treatment complications e.g. patients with a hypersensitivity to tildrakizumab, abiraterone, prednisolone, or any of the drug excipients.
25. Patients with female partners of child-bearing potential (unless they agree to take measures not to father children by using a barrier method of contraception [condom plus spermicide] or to sexual abstinence effective from the first administration of any of the study drugs throughout the trial and for six months afterwards. Men with partners of child-bearing potential must also be willing to ensure that their partner uses an effective method of contraception for the same duration for example, hormonal contraception, intrauterine device, diaphragm with spermicidal gel or sexual abstinence). Men with pregnant or lactating partners must be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure of the foetus or neonate.

    NB. Abstinence is only considered to be an acceptable method of contraception when this is in line with the preferred and usual lifestyle of the participants. Periodic abstinence (e.g., calendar, ovulation, sympathothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
26. Prior bone marrow transplant.
27. Extensive radiotherapy to greater than 25% of bone marrow within 8 weeks.
28. Any other condition, which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
29. Symptoms of COVID-19 and/or documented COVID-19 infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Phase I - To describe the safety and tolerability of abiraterone acetate and tildrakizumab when given in combination. To establish a RP2D for tildrakizumab, in combination with abiraterone. | 20 months
  To determine a maximum tolerated dose (MTD) of tildrakizumab by establishing the dose at which the DLT rate is as close to the target DLT rate of 15% as possible, in combination with abiraterone at 500 mg OD with prednisolone at 5 mg bid, and is deemed to be tolerable by the Safety Review Committee. This will be the RP2D for tildrakizumab.
Phase II - To determine the antitumour activity of tildrakizumab (at RP2D) in combination with abiraterone in men with mCRPC. | 12 months
  Antitumour activity will be defined by response rate on the basis of the following outcomes. If any of the following occur, patients will be considered to have responded:
  * PSA decline ≥ 50% criteria confirmed 4-weeks or later and/or,
  * Confirmed soft tissue objective response by RECIST (v1.1) in patients with measurable disease and/or,
  * ONLY for patients with detectable circulating tumour cell (CTC) count of ≥ 5/7.5ml blood at baseline, conversion of CTC count to <5/7.5ml blood nadir.

SECONDARY OUTCOMES:
Phase I - To investigate the PD effects of the tildrakizumab and abiraterone combination in men with mCRPC. | 20 months
  Measuring the impact of the downregulation of IL-23 signaling in tumour, also evaluating the downregulation of androgen receptor (AR), AR splice variants, and AR target genes.
Phase I - To characterize the PK profile of the tildrakizumab and abiraterone combination in men with mCRPC - CMax. | 20 months
  Determine peak plasma concentration (Cmax) of tildrakizumab and abiraterone when dosed together.
Phase I - To characterize the PK profile of the tildrakizumab and abiraterone combination in men with mCRPC - T1⁄2. | 20 months
  Determine the terminal elimination half-life (T1⁄2) of tildrakizumab and abiraterone when dosed together.
Phase I - To characterize the PK profile of the tildrakizumab and abiraterone combination in men with mCRPC - AUC | 20 months
  Determine the area under the plasma concentration versus time curve (AUC) of tildrakizumab and abiraterone when dosed together.
Phase I - To identify molecular determinants of response and anti-tumour activity of the combination of tildrakizumab and abiraterone in men with mCRPC. | 20 months
  Determine biomarkers of response, including but not limited to PTEN loss, MYC amplification, and intra-tumour MDSC counts, in tumour biopsies from responders and non-responders.
Phase I - To determine preliminary anti-tumour activity of the tildrakizumab and abiraterone combination in men with mCRPC. | 20 months
  Response and progression will be determined using the same measures as that described for the primary objective of the Phase II study.
Phase I - To evaluate progression-free survival (PFS) in mCRPC patients receiving the tildrakizumab and abiraterone combination. | 20 months
  PFS will be measured from the date of addition of tildrakizumab to abiraterone to the date of progression as determined by radiological criteria (RECIST v 1.1, PCWG3 bone scan criteria) or unequivocal clinical progression necessitating drug discontinuation (e.g. worsening pain, spinal cord compression, need for other anticancer therapy).
Phase I - To estimate the OS in mCRPC patients receiving the combination of tildrakizumab and abiraterone. | 20 months
  OS will be measured from the date of addition of tildrakizumab to abiraterone to the date of death (whatever cause).
Phase II - To evaluate PFS in mCRPC patients receiving the tildrakizumab and abiraterone combination. | 12 months
  PFS will be measured from the date of addition of tildrakizumab to abiraterone to the date of progression as determined by radiological criteria (RECIST v 1.1, PCWG3 bone scan criteria) or unequivocal clinical progression necessitating drug discontinuation (e.g. worsening pain, spinal cord compression, need for other anticancer therapy).
Phase II - To estimate the biochemical anti-tumour activity of tildrakizumab and abiraterone in mCRPC patients - time to PSA progression. | 12 months
  The time to PSA Progression will be measured from the date of addition of tildrakizumab to abiraterone.
Phase II - To estimate the biochemical anti-tumour activity of tildrakizumab and abiraterone in mCRPC patients - duration of PSA decline by ≥ 50%. | 12 months
  The duration of PSA decline by ≥ 50%, where this is seen in responding patients.
Phase II - To estimate the biochemical anti-tumour activity of tildrakizumab and abiraterone in mCRPC patients - maximum PSA decline. | 12 months
  The maximum PSA decline experienced per patient. This will be measured following the addition of tildrakizumab to abiraterone.
Phase II - To estimate the biochemical anti-tumour activity of tildrakizumab and abiraterone in mCRPC patients - maximum percentage of PSA decline. | 12 months
  The maximum percentage of PSA decline experienced per patient. This will be measured following the addition of tildrakizumab to abiraterone.
Phase II - To determine the pattern of radiologic response to tildrakizumab and abiraterone in mCRPC patients. | 12 months
  Time to radiological progression (RECIST 1.1 & PCWG3 Bone Scan criteria). Radiologic PFS (rPFS).
Phase II - To identify molecular determinants of response and anti-tumour activity of the combination of tildrakizumab and abiraterone in men with mCRPC. | 12 months
  Determine biomarkers of response, including but not limited to PTEN loss, MYC amplification, and intra-tumour MDSC counts, in tumour biopsies from responders and non-responders.
Phase II - To further investigate the PD effects of the tildrakizumab and abiraterone combination in men with mCRPC. | 12 months
  Measure the impact of the downregulation of IL-23 signaling in tumour, also evaluating the downregulation of androgen receptor (AR), AR splice variants, and AR target genes
Phase II - To determine the rate of response based on CTC conversion. | 12 months
  Rate of CTC conversion from ≥ 5/7.5 ml blood to < 5/7.5 ml
Phase II - To estimate the OS in mCRPC patients receiving the combination of tildrakizumab and abiraterone. | 12 months
  OS will be measured from the date of addition of tildrakizumab to abiraterone to the date of death (whatever cause).
Phase II - To further characterise the safety and tolerability profile of the combination of tildrakizumab and abiraterone in men with mCRPC. | 12 months
  Causality and grading severity of each adverse event related to the tildrakizumab and abiraterone combination according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0

OTHER OUTCOMES:
To determine mechanisms of resistance to the combination of tildrakizumab and abiraterone. | 32 months
  Deregulation, amongst others, of IL-23, STAT proteins, AR, AR splice variants.
To assess putative predictive biomarkers of response to this combination. | 32 months
  Correlate anti-tumour activity of the combination of tildrakizumab and abiraterone with the detection of putative predictive biomarkers of response and resistance in archival tumours, paired fresh tumour biopsies, and plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Johann De Bono, MD, Study Director — National Health Service, United Kingdom
Locations (6):
- Bellinzona Hospital, Bellinzona, Switzerland
- United Kingdom (5):
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Belfast City Hospital, Belfast, UK
  - The Royal Marsden Hospital Foundation Trust, Sutton, UK
  - Addenbrooke's Hospital, Cambridge
  - University Hospitals Southampton NHS Foundation Trust, Southampton